CLINICAL TRIAL: NCT05009680
Title: GULLIVER-2 - A Single (Open-label) and Repeat Dose (Randomised, Placebo-controlled) Trial to Assess the Safety, Tolerability and Pharmacokinetics of GB1211 in Participants With Hepatic Impairment (Child Pugh B & C)
Brief Title: A Single and Repeat Dose Trial in Participants With Hepatic Impairment
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Galecto Biotech AB (Industry)
Collaborators: Comac Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GULLIVER-2
Record Dates: First submitted 2021-07-27; First posted 2021-08-17 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-02

CONDITIONS: Hepatic Impairment
Keywords: Child Pugh B; Child Pugh C; Liver Cirrhosis; Galectin 3 Inhibitor
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Intervention Model Description: Parts 1 & 3 Open Label, Single Dose Part 2 Randomised to either GB1211 or Placebo
Who Masked: Participant
Masking Description: Parts 1 & 3 - Open Label, Single Dose Part 2 - Double-blind. The blinding will be maintained throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Part 1 GB1211, Single Dose (Child Pugh B) (Experimental): GB1211 is a galectin-3 inhibitor an orally available small molecule anti-fibrotic. It is administered orally twice a day.
  Interventions: Drug: GB1211
- Part 1 GB1211 Healthy Matched Participants, Single Dose (Experimental): GB1211 is a galectin-3 inhibitor an orally available small molecule anti-fibrotic. It is administered orally twice a day.
  Interventions: Drug: GB1211
- Part 2 GB1211 Multiple Dose, Twice a day (Child Pugh B) (Experimental): GB1211 is a galectin-3 inhibitor an orally available small molecule anti-fibrotic. It is administered orally twice a day.
  Interventions: Drug: GB1211
- Part 2 Placebo, Twice a day (Child Pugh B) (Placebo Comparator): Placebo is administered twice daily
  Interventions: Drug: Placebo
- Part 1 GB1211, Single Dose (Child Pugh C) (Experimental): Part 1 GB1211 Healthy Matched Participants, Single Dose
  Interventions: Drug: GB1211
- Part 3 GB1211 Healthy Matched Participants, Single Dose (Experimental): Part 1 GB1211 Healthy Matched Participants, Single Dose
  Interventions: Drug: GB1211

INTERVENTIONS:
Drug: GB1211 — GB1211 is a galectin-3 inhibitor an orally available small molecule anti-fibrotic. It is administered orally twice a day
  Arms: Part 1 GB1211 Healthy Matched Participants, Single Dose; Part 1 GB1211, Single Dose (Child Pugh B); Part 1 GB1211, Single Dose (Child Pugh C); Part 2 GB1211 Multiple Dose, Twice a day (Child Pugh B); Part 3 GB1211 Healthy Matched Participants, Single Dose
Drug: Placebo — Placebo is administered orally twice a day
  Arms: Part 2 Placebo, Twice a day (Child Pugh B)

SUMMARY:
This study is a a single (open-label) and repeat dose (randomised, placebo controlled) trial to assess the safety, tolerability and pharmacokinetics of GB1211 (Gal-3 inhibitor) in participants with hepatic impairment (Child Pugh B and Child Pugh C)

DETAILED DESCRIPTION:
PART 1 A single dose, open-label safety and PK study of GB1211 administered to participants with moderate hepatic impairment (Child Pugh B) and to matched healthy participants (controls).

PART 2 A randomised, double-blind, placebo-controlled study in participants with moderate hepatic impairment (Child Pugh B). GB1211 or placebo will be administered daily for 12 weeks.

PART 3 A single dose, open-label safety and PK study of GB1211 administered to participants with severe hepatic impairment (Child Pugh C) and to healthy participants (controls).

ELIGIBILITY:
Inclusion Criteria:

Main Inclusion Criteria:

1. Males or females, of any race, ≥ 18 and ≤ 75 years of age at enrolment
2. Body mass index (BMI) of ≥ 18-40 kg/m2
3. Participants with hepatic impairment:

   1. PART 1 and PART 2: Moderate hepatic impairment, as defined by the Child-Pugh score (Child-Pugh B) [1] who exhibit physical signs consistent with stable hepatic impairment and free of significant medical disorders unrelated to their hepatic disorder and are on stable concomitant medication for 2 weeks prior to and for the duration of this study
   2. PART 3: Severe hepatic impairment as defined by the Child-Pugh score (Child Pugh C) who exhibit physical signs consistent with stable hepatic impairment and free of significant medical disorders unrelated to their hepatic disorder and are on stable concomitant medication for 2 weeks prior to and for the duration of this study
4. Healthy participants (controls) in PART 1 and PART 3:

   1. Healthy as determined by the investigator, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac assessment
   2. Match at least one of the participants with moderate or severe hepatic impairment with respect to gender, age (±10 years), and body mass index (BMI) ± 15% (ensure every participant with hepatic impairment has at least 1 matched control)
5. Women of non-childbearing potential defined as permanently sterile or postmenopausal
6. Males will agree to use contraception throughout the study and until 90-days after the Follow-up visit
7. Male participants must agree to refrain from sperm donation from the date of Randomisation (Day 1) until 90 days after the Follow up visit
8. Able to comprehend and willing to sign an ICF and to abide by the study restrictions

Exclusion Criteria:

All parts and all groups (control healthy volunteers and hepatic impairment)

1. History of an organ transplant, including a remote history of bone marrow transplant
2. History of febrile illness within 7 days prior to the first dose of study drug or participants with evidence of active infection
3. Use of any oral glucocorticoids at any dose within 30 days prior to Screening and until study completion
4. Have previously completed or withdrawn from a study investigating GB1211 and have previously received the investigational product
5. Participant who, in the opinion of the Investigator (or Designee), should not participate in this study
6. Vulnerable/institutionalised patients
7. Patients related to Principal Investigator (PI)/site staff
8. If female, the participant is of child-bearing potential
9. Participation in a clinical study involving administration of an investigational agent e.g. new chemical entity or a biological product in the past 90 days (or 5 multiples of half-life, whichever is longer) prior to dosing.
10. Medical history of cardiac disease and/or clinically significant ECG abnormalities. An abnormal ECG is defined as PR > 220 msec, QRS complex >120 msec, QTcF > 450 msec (males) and > 470msec (females), or any other morphological changes, other than nonspecific T-wave changes
11. Donation or loss of ≥ 400 mL blood or plasma less than 4 weeks prior to screening, or longer if required by local regulations
12. Positive HIV test
13. Have received live vaccine(s) within 30 days prior to Screening or who will require a vaccine(s) and until study completion
14. Use of any medications/products that may inhibit biliary excretion, e.g. bile salt chelators, mycophenolic acid, warfarin, and digoxin, within 30 days prior to Screening and until study completion
15. Use of any medications/products that may inhibit renal excretion; e.g. cimetidine, pyrimethamine, dolutegravir, probenecid, within 30 days prior to Screening and until study completion
16. Use of any medications/products that are known inhibitors of P-gp (e.g. clarithromycin, fostamatinib, quinidine, quinine) and inducers of P-gp (e.g. carbmazepine, rifampin, St. John's wort) within 30 days prior to Screening and until study completion

    Additional exclusion criteria for matched healthy control subjects:
17. Use of any prescription or non-prescription medication (OTC), herbal medication, dietary supplements or vitamins during 30 days prior to dosing. Acetaminophen is acceptable
18. History or presence of liver disease or liver injury as indicated by an abnormal liver function profile such as AST, ALT, alkaline phosphatase, or serum bilirubin
19. A positive Hepatitis C test or a positive Hepatitis B surface antigen (HBsAg)
20. Estimated glomerular filtration rate (eGFR) < 80 mL/[min*1.73 m²] (estimated using the Modification of Diet in Renal Disease [MDRD] equation) at Screening

    Additional exclusion criteria for hepatic impaired subjects:

    Participants meeting any of the following exclusion criteria are not to be enrolled in the study/randomised to treatment:
21. History of any known serious disease (such as cancer, except skin basal cell carcinomas, major infection, clinically significant gastrointestinal disorder, major autoimmune disease) or other disease which in the Investigator's opinion would exclude the patient from the study
22. Estimated glomerular filtration rate (eGFR) < 40 mL/[min*1.73 m²] (estimated using the [MDRD] equation) at Screening
23. Use of any hepatotoxic drug (e.g. methotrexate, isoniazid, amiodarone) within 30 days of Screening and until study completion
24. Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's Wort, or other putatively hepatoprotective herbal remedies such as milk thistle derivatives, within 30 days prior to dosing, unless deemed acceptable by the Investigator (or Designee). Milk thistle derivates or other hepatoprotective herbal remedies are allowed if stable dose is administered 30 days before dosing
25. Use or intend to use slow release medications/products considered to still be active within 14 days prior to Randomisation, unless deemed acceptable by the Investigator (or Designee)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-09-09 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2023-07-04 (Estimated)

PRIMARY OUTCOMES:
Parts 1 Safety and Tolerability of GB1211 | 11 Days
  Incidence and severity of adverse events as reported by investigators
Parts 2 Safety and Tolerability of GB1211 | 12 Weeks
  Incidence and severity of adverse events as reported by investigators
Parts 3 Safety and Tolerability of GB1211 | 11 Days
  Incidence and severity of adverse events as reported by investigators

SECONDARY OUTCOMES:
Part 2 Collagen Production and Breakdown Biomarkers | 12 Weeks
  Assessment of liver fibrosis using pro-C3, CK18 and PAI-1 Biomarkers
Part 2 Changes on liver and spleen stiffness | 12 Weeks
  Assessment of liver and spleen stiffness measured by vibration control transient elastography
Part 2 Changes in Liver Functional Capacity | 12 Weeks
  Assessment of Liver functional Capacity measured by 13C methacetin breath test

CONTACTS AND LOCATIONS:
Overall Officials: Zahariy Krastev, MD, Principal Investigator — Comac Medical
Locations (4):
- Bulgaria (4):
  - COAMC Medical, Sofia
  - Gastroenterology Clinic, Lozenets district, Sofia
  - Diagnostic-Advisory center 'ALEKSANDROVSKA" Ltd, Sofia
  - University Multiprofile Hospital, Clinic of gastroenterology, Sofia, Оborishte District

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aslanis V, Gray M, Slack RJ, Zetterberg FR, Tonev D, Phung D, Smith B, Jacoby B, Schambye H, Krastev Z, Ungell AL, Lindmark B. Single-Dose Pharmacokinetics and Safety of the Oral Galectin-3 Inhibitor, Selvigaltin (GB1211), in Participants with Hepatic Impairment. Clin Drug Investig. 2024 Oct;44(10):773-787. doi: 10.1007/s40261-024-01395-7. Epub 2024 Oct 2. PMID 39358661